CLINICAL TRIAL: NCT05311631
Title: Breastfeeding - a Good Start Together
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Committee for Health Education (Other); 21 municipalities in Denmark (Unknown); Nordea-fonden (Unknown); Det Obelske Familiefond (Unknown)
Responsible Party: Principal Investigator, Sarah Fredsted Villadsen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Breastfeeding
Record Dates: First submitted 2022-03-11; First posted 2022-04-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive
Keywords: Social inequality; Breastfeeding self-efficacy; Breastfeeding support; Complex interventions; Public health
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Clusters (municipalities) are randomized to either intervention or control (standard care). Intervention coverage 6000 infants and their families in intervention municipalities. Primary trial outcome is assessed using survey data where 3339 families from the intervention and control arm will be enrolled according to the power calculation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Improved breastfeeding support provided by health visitors supporting families after discharge from maternity ward at hospital. The intervention is implemented into the existing national health visitor program that is offered free of charge to all. The program is accepted by more than 95% of families.
  Interventions: Behavioral: Breastfeeding support
- Control (No Intervention): Health visitors in the control municipalities will give breastfeeding support according to standard care.

INTERVENTIONS:
Behavioral: Breastfeeding support — The core of the intervention is a trustful relation between the health visitor and the families based on principles of needs based communication. Health visitors will enhance parents' action competence based on breastfeeding self-efficacy, focusing on parents' wishes and needs.
  The breastfeeding support includes four main messages: joint parenting task, skin-to-skin contact, frequent breastfeeding, and good positioning.
  Training of health visitors includes e-learning and a two-day course with physical attendance. Supportive materials are developed including communicative support tools and a web-page providing support and knowledge when the health visitor is off hours.
  All families in intervention sites accepting the health visitor program will receive the improved breastfeeding support. Families in the high-risk group are offered an intensified intervention with close follow-up by telephone in planned time-intervals, thus a higher dose of the intervention.
  Arms: Intervention

SUMMARY:
The Breastfeeding - a Good Start Together intervention study aims to increase the proportion of women who breastfeed for four and six months, and proportionately more in a group of women who are in risk of early breastfeeding cessation; and thus reduce social inequality of mother and infant health.

DETAILED DESCRIPTION:
Breastfeeding has numerous health benefits for both mothers and children, and the World Health Organization recommends exclusive breastfeeding for six months. Still, only 12 % of mothers in Denmark breastfeed exclusively at six months postpartum and breastfeeding is subject to significant social inequality. Mothers of young age (below 25 years) and with low educational attainment (not exceeding primary school or vocational) breastfeed for a shorter duration of time than their counterparts. Thus, this group is in high risk of early breastfeeding cessation and is hereafter termed 'the high-risk group'.

The Breastfeeding - a Good Start Together intervention consists of theory based breastfeeding support, supported by printed materials and a web-page providing support and knowledge for families when health visitors are off work, and an intensified intervention aimed at the high-risk group, comprising close follow-up by telephone and an extra home visit. In total, the high-risk group will receive seven telephone calls during week two post partum and 15 weeks post partum, with the highest intensity in the first month (contact once a week), gradually decreasing as the child grows older (contact every second week during the second month, and every third week during the third and fourth month).

Hypothesis: Improving the relationship between health visitors and new families, drawing on tailoring of the communication, which ensures that breastfeeding support matches the needs of the family, will enhance trust and therefore the likelihood of families reaching out to the health nurse when breastfeeding problems occur and thus improving chances of successful breastfeeding in a longer duration of time. Moreover, the theory based breastfeeding support will make the support more easily attainable for families, independent of their sociodemographic background. Improving chances of a successful breastfeeding will improve mother and infant health, the latter especially with regards to lower infant morbidity related to nutrition.

The intervention is a complex intervention, designed as a cluster-randomized trial. Twenty-one municipalities situated in the North Denmark Region and Region of Southern Denmark participate in the study, and according to the number of births among inhabitants these have been randomized to either intervention or control group; 11 intervention municipalities and 10 control municipalities. Basing the randomization on number of births proved to successfully account for other factors, such as rural or urban areas and proportion of high-risk individuals.

The intervention will be implemented from March 2022-December 2023, with data collection commencing April 2022. Health visitors in the intervention municipalities will receive training before delivering the new breastfeeding counselling to the families. The training is expected to reach 225 health visitors in the intervention municipalities and 6000 families of whom 30-40% are in the high-risk group. After the trial period, health visitors in the control municipalities will receive the same training.

The primary outcome measures of the intervention is breastfeeding duration and proxies for infant morbidity related to nutrition. Secondary outcomes are the families' perception of their relationship with the health visitor and parents' action competence and self-efficacy related to breastfeeding.

The primary and secondary outcome measures, are studied in a survey study using electronic questionnaires distributed to mothers recruited through the health-visiting programme at three time-points, and to fathers/partners at one time-point. Further, the effectiveness of the intervention will be analysed using register-data. A difference-in-difference design is applied to measure changes in primary outcomes from before to after the intervention period in both intervention sites and control sites.

The overall target group of the intervention study is all new families accepting the health visiting program with a specific high-risk group of families with mothers of young age or who have low educational attainment. Outcomes of the trial will be analysed for the total population and for the sub-group.

For sample size calculation an estimation of 8 clusters in the intervention arm and 8 clusters in the control arm were used, as this calculation was made prior to successfully recruiting a total of 21 clusters to the trial. The investigators expect a participation of 80% with an attrition of 30%. The ambition is to improve the breastfeeding duration in the intervention clusters to the national level, corresponding to an OR 1.32. With an interclass correlation coefficient of 0.001, a strength of 80% and a 5% significance level can be reached if data are collected from 111 mothers in each cluster, including 52 mothers from the high-risk group in each cluster.

All effectiveness analyses will be using an intention-to-treat approach and will account for the clustering of individuals and potential confounding in a controlled mixed effect regression.

The implementation of the intervention will be analysed in a process evaluation using qualitative and quantitative data. A realist evaluation using qualitative data will explore the mechanisms of change in the intervention, and will highlight what works for whom, under what circumstances.

Further, a health economic evaluation will be performed as a cost-effectiveness analysis where health benefits are measured as changes in the proportion of women breastfeeding at four months post partum, and as a cost-utility analysis where health benefits are measured as gained Quality Adjusted Life-Years (QALYs). Moreover, an analysis of the costs of the intervention related to the costs (and possible savings) in the health system surrounding the intervention sites.

ELIGIBILITY:
Inclusion Criteria:

1a. Families discharged <72 hours post partum (from 26 April 2022 - 17 January 2023)

1b. Families discharged < 7 days post partum (from 18 January 2023 onwards due to lower than expected recruitment rate)

2. Families with intention of breastfeeding

Exclusion Criteria:

* Insufficient skills in Danish or English language to be able to answer questionnaires and understand interventions conveyed in Danish or English
* Families with mothers with known substance abuse or addiction
* Families expecting more than one child
* Families having delivered preterm, prior to 37 weeks of gestation
* Families with mothers or child having difficulty breastfeeding due to a known morbidity or disablement

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5010 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal self-report of breastfeeding status (full vs not full) | Four months post partum
  Self-reported breastfeeding measured in questionnaires by the mothers and health visitors' record of breastfeeding status. Full breastfeeding is conceptualized as exclusive breastmilk-feeding after discharge from the hospital. In Denmark, the concept allows for a supplement to mother's milk of water and the like and / or a maximum of one meal with infant formula per week.

SECONDARY OUTCOMES:
Maternal self-report of breastfeeding status (full vs not full) | Six months post partum
  Self-reported breastfeeding measured in questionnaires by the mother. In Denmark, full breastfeeding allows for a supplement to mother's milk of water and the like and / or a maximum of one meal with infant formula per week
Infant thriving - jaundice | From birth to one months post partum
  Change in readmissions of children dur to jaundice is used as an indicator of infant morbidity related to nutritional problems. Measured by self-report in questionnaires and obtained from Danish registers of hospital admissions.
Infant thriving - weight loss | From birth to one months post partum
  Change in readmissions of children due to weight loss is used as an indicator of infant morbidity related to nutritional problems. Measured by self-report in questionnaires and obtained from Danish registers of hospital admissions.
Infant thriving - dehydration | From birth to one months post partum
  Change in readmissions of children due dehydration is used as an indicator of infant morbidity related to nutritional problems. Measured by self-report in questionnaires and obtained from Danish registers of hospital admissions.
Breastfeeding problems | One week and one month post partum
  Change in frequency of pain during breastfeeding, sores or cracks on nipples, problems with latching on, the experience of having too little milk, the experience of having too much milk, the experience that the infant wants to feed very frequently, the experience of long duration of each breastfeeding, problems with low infant weight gain, breast tension, mastitis. This will be assessed through maternal self report in questionnaires.
Trust in visiting nurse | One month and four months
  Maternal self reported feeling of being seen, respected and heard
Breastfeeding self-efficacy | One month
  Maternal and paternal self report in survey
Duration of full breastfeeding (weeks) | From birth to six months postpartum
  Self-reported full breastfeeding measured in questionnaires by the mothers.
Any breastfeeding | From birth to 12 months postpartum
  Self-reported breastfeeding status measured in questionnaires by the mothers. Any breastfeeding includes a mothers report of some to full breastfeeding.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid SM Nilsson, PhD, Principal Investigator — The Danish Committee of Health Education
Locations (21):
- Denmark (21):
  - Aabenraa Kommune, Aabenraa
  - Jammerbugt Kommune, Aabybro
  - Vesthimmerland Kommune, Aars
  - Assens Kommune, Assens
  - Billund Kommune, Billund
  - Esbjerg Kommune, Esbjerg
  - Fredericia Kommune, Fredericia
  - Frederikshavn Kommune, Frederikshavn
  - Haderslev Kommune, Haderslev
  - Mariagerfjord Kommune, Hobro
  - Kolding Kommune, Kolding
  - Middelfart Kommune, Middelfart
  - Morsø Kommune, Nykøbing Mors
  - Odense Kommune, Odense
  - Faaborg-Midtfyn Kommune, Ringe
  - Svendborg Kommune, Svendborg
  - Sønderborg Kommune, Sønderborg
  - Thisted Kommune, Thisted
  - Tønder Kommune, Tønder
  - Varde Kommune, Varde
  - Vejen Kommune, Vejen Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobsen MH, Gadeberg AK, Rossau HK, Nilsson IMS, Villadsen SF. Understanding fathers' responses to breastfeeding as a "shared parental task": a realist evaluation of a Danish breastfeeding support intervention. Arch Public Health. 2025 Nov 27;83(1):299. doi: 10.1186/s13690-025-01790-2. PMID 41299756
- [Derived] Rossau HK, Gadeberg AK, Strandberg-Larsen K, Nilsson IMS, Villadsen SF. Process evaluation of a breastfeeding support intervention to promote exclusive breastfeeding and reduce social inequity: a mixed-methods study in a cluster-randomised trial. Int J Equity Health. 2024 Oct 8;23(1):204. doi: 10.1186/s12939-024-02295-0. PMID 39380053
- [Derived] Nilsson I, Busck-Rasmussen M, Villadsen SF. Development of a complex intervention to strengthen municipality-based breastfeeding support to reduced social inequity in breastfeeding. Arch Public Health. 2024 Oct 2;82(1):174. doi: 10.1186/s13690-024-01401-6. PMID 39358759
- [Derived] Rossau HK, Nilsson IMS, Gadeberg AK, Forman JL, Strandberg-Larsen K, Nielsen J, Villadsen SF. Strengthening health visitors' breastfeeding support: Results from a cluster randomised study. Nurse Educ Pract. 2024 Jul;78:104033. doi: 10.1016/j.nepr.2024.104033. Epub 2024 Jun 18. PMID 38905959
- [Derived] Rossau HK, Nilsson IMS, Busck-Rasmussen M, Ekstrom CT, Gadeberg AK, Hirani JC, Strandberg-Larsen K, Villadsen SF. Effectiveness of a community-based support programme to reduce social inequality in exclusive breastfeeding: study protocol for a cluster-randomised trial. BMC Public Health. 2023 Mar 8;23(1):450. doi: 10.1186/s12889-023-15256-z. PMID 36890478